CLINICAL TRIAL: NCT01738178
Title: Caffeine as a Therapeutic Agent in Parkinson's Disease
Brief Title: Caffeine as a Therapy for Parkinson's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Pontifícia Universidade Católica do Paraná (Other); University of Calgary (Other); University of Newfoundland and Eastern Health (Unknown); University Health Network, Toronto (Other); UBC Hospital (Unknown); Movement Disorder Clinic - Deer Lodge Centre (Unknown); The Ottawa Hospital (Other)
Responsible Party: Principal Investigator, Ron Postuma, Neurologist, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2778
Record Dates: First submitted 2012-11-28; First posted 2012-11-30 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control - Placebo (Placebo Comparator): These participants will receive placebo tablets during the first 5 years
  Interventions: Drug: Placebo
- Caffeine group (Active Comparator): This group of participants will receive caffeine tablets.
  Interventions: Drug: Caffeine

INTERVENTIONS:
Drug: Caffeine
  Arms: Caffeine group
Drug: Placebo
  Arms: Control - Placebo

SUMMARY:
Parkinson's disease is a common neurodegenerative disorder in which patients experience progressive motor disability and many disabling non-motor symptoms. Recent studies have consistently found that people who do not use caffeine are at higher risk of developing Parkinson's disease. This suggests that caffeine may have potential as a treatment for PD.

In a pilot study of caffeine for daytime sleepiness in PD, there was evident benefit on the motor manifestations of disease. There have been other lines of evidence that have suggested caffeine could be useful in PD. This study is to evaluate the efficacy of caffeine 200 mg BID vs matching placebo for motor and non-motor aspects of disease. This will be in three stages. In the first six-month stage, medications will be held constant, to see whether caffeine does have motor benefits. Then we will perform a four-year extension stage to define if the effects of caffeine persist (or even magnify), and to see if caffeine helps reduce dose of other PD meds and/or prevents their side effects. Finally, we will finish with a six-month stage in which we will place all patients on caffeine - this will allow us to assess caffeine's use in later disease, but more importantly, will assess whether early use of caffeine produces long term changes beyond its immediate effects.

ELIGIBILITY:
Inclusion Criteria:

All patients must have idiopathic PD diagnosed as parkinsonism according to the UK brain bank criteria, and PD considered the likeliest underlying cause according to the treating physician. Other inclusion criteria include:

1. PD diagnosis: between 6 months and 8 years
2. Hoehn and Yahr stage I-III
3. Age at least 45 and less than 75 (to optimize survival over the 5-year trial).
4. Receiving symptomatic therapy for PD for at least 6 months. Dose must have been stable over the previous 3 months.

Exclusion Criteria:

1. Caffeine intake >150 mg per day (i.e. more than one cup of filtered coffee per day) or prescribed adenosine antagonists - caffeine intake will be measured by a standardized intake questionnaire. Intake will be converted into estimated caffeine mg dose by standard caffeine-content charts.
2. Active peptic ulcer disease, or symptomatic gastroesophageal reflux disease.
3. Supraventricular cardiac arrhythmia (such as atrial fibrillation or atrial flutter) - Electrocardiogram will be measured at baseline to rule out supraventricular tachycardia.
4. Uncontrolled hypertension - systolic bp >170 or diastolic bp >110 on two readings.
5. Pre-menopausal women who are not using effective methods of birth control
6. Cognitive impairment, defined as MoCA <23/30.
7. Moderate-Severe Depression, as defined by a Beck Depression Inventory score of >19.
8. Changes to antiparkinsonian medication in the last 3 months, or changes to antiparkinsonian medication are anticipated during the next six months.
9. Current use of lithium or clozapine (pharmacokinetic interactions).

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2014-04; Primary Completion 2016-05-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Motor manifestations associated with Parkinson's disease | every 6 months
  For each stage of the study, the MDS-Unified Parkinson Disease Rating Scale (MDS-UPDRS)will be used as the primary outcome. The MDS-UPDRS is the standard scale used for grading severity of PD - its revised 2008 version has more standardized motor assessment, better sensitivity to change in early-mid stages, and a broader assessment of non-motor PD. It starts with a patient self-administered questionnaire covering activities of daily living, motor symptoms, and non-motor domains. There is then a scored clinical interview assessing cognitive and psychiatric symptoms and motor complications. The Hoehn and Yahr scale (5-point overall disease severity index) is included3. Finally, there is a formal examination component (Part III) (performed in the medication 'on' state for this study).

SECONDARY OUTCOMES:
MDS-UPDRS components and subscales - each individual component will be assessed, including: | every 6 months
  1. motor symptoms, according to each subscale question. These include speech deficits, swallowing dysfunction, motor activities of daily living (dressing, feeding, turns in bed, etc), tremor, gait slowing, freezing, and falls
  2. non-motor symptoms, according to each subscale question. These include constipation, urinary dysfunction, sexual dysfunction, orthostatic symptoms, depression, anxiety, cognitive symptoms, apathy, somnolence, insomnia, pain, and fatigue.
  3. motor complications - motor fluctuations and dyskinesia
  4. Hoehn and Yahr staging (a five-point global staging system for PD).
Cognition | every 6 months
  Although cognitive symptoms are addressed with the UPRDS, we will include two objective measures, the Montreal Cognitive Assessment (MoCA), and Mini-mental State Examination. The MoCA is a brief cognitive test, which is used extensively in PD. The MMSE will be used in diagnosis of dementia. Dementia will be assessed according to Level I MDS criteria. ADL impairment due to cognitive loss will be documented according to MDS criteria.
Sleep | every 6 motnhs
  Because caffeine may have special effectiveness for sleep disorders, we will include additional sleep questionnaires, including
  1. the SCOPA-sleep8 nighttime scale.
  2. the SCOPA-sleep8 daytime scale
  3. the REM sleep behavior disorder single-question screen (RBD1Q)
Quality of life | every 6 months
  The Parkinson's Disease Questionnaire-8 is a quality of life index for PD with 8 self-administered items assessing motor function, gait, mood, cognition, etc.
Medication utilization | evry 6 months
  To assess caffeine's potential medication-sparing benefit, we will quantify all medications at each visit. Levodopa-dose equivalents will be calculated with standard criteria. Total medication cost will be calculated using current Canadian pharmacy pricing.
Tolerability and side effects of caffeine | every 6 motnhs
  A structured questionnaire will screen for irritability, symptoms of gastrointestinal reflux, diarrhea, sleepiness, palpitations, sweating, and tremulousness. In addition, open-ended questions will allow reporting of other side effects. Blood pressure will be measured at each visit to exclude new-onset hypertension, and orthostatic hypotension will be objective assessed with blood pressure measurements lying and standing (1 minute).

CONTACTS AND LOCATIONS:
Overall Officials: Ronald B Postuma, MD, MSc, Principal Investigator — Research Insitute of the MUHC
Locations (8):
- Parana Parkinson Association - Pontifical Catholic University of Parana, Curitiba, Paraná, Brazil
- Canada (7):
  - Heritage Medical Research Clinic - University of Calgary, Calgary, Alberta
  - UBC Hospital - Pacific Parkinson's Research Centre, Vancouver, British Columbia
  - Movement Disorder Clinic - Deer Lodge Centre, Winnipeg, Manitoba
  - Memorial University of Newfoundland, St. John's, Newfoundland and Labrador
  - The Ottawa Hospital - Civic Campus, Ottawa, Ontario
  - Toronto western Hospital - Movement Disorders Research Centre, Toronto, Ontario
  - McGill University Health Center, Montreal, Quebec

REFERENCES:
- [Derived] Postuma RB, Anang J, Pelletier A, Joseph L, Moscovich M, Grimes D, Furtado S, Munhoz RP, Appel-Cresswell S, Moro A, Borys A, Hobson D, Lang AE. Caffeine as symptomatic treatment for Parkinson disease (Cafe-PD): A randomized trial. Neurology. 2017 Oct 24;89(17):1795-1803. doi: 10.1212/WNL.0000000000004568. Epub 2017 Sep 27. PMID 28954882